CLINICAL TRIAL: NCT05089747
Title: MAster Protocol Studying the Impact of Blood Biopsy on Screening, Diagnosis, Diagnostic and Follow-up of Solid Cancer in Adult
Brief Title: CIRculating CANcer MAster-Protocol
Acronym: CIRCAN MAP
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0918
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Adult With Solid Cancer
Keywords: liquid biopsy; solid cancer
MeSH Terms: interventions — Blood Specimen Collection; MicroRNAs; Cell-Free Nucleic Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult with solid cancer. No intervention.
  Interventions: Biological: Blood sampling for biomarker analysis (microRNA, circulating DNA…)

INTERVENTIONS:
Biological: Blood sampling for biomarker analysis (microRNA, circulating DNA…) — From one to four blood samplings: at diagnosis, after the first cycle of treatment, end of treatment, progressive disease (or end of study).

SUMMARY:
This exploratory study will focus on the development of the analyses of blood biomarkers to better understand the circulating biomarkers associated with cancer diagnosis, treatment efficacy and progressive disease

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18y)
* Owing a social security insurance
* Any solid cancer diagnosed by histopathology or cytology
* Patient with blood sampling required as per standard of care
* Informed consent signed

Exclusion Criteria:

* Refusal to participate
* No blood sampling required as per standard of care
* Hemoglobin < 7g/dl (< 9g/dl if respiratory or cardiovascular disease history)
* Heterologous blood transfusion in the last 48 hours
* Weight under 20 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with solid cancer
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2047-12-01 (Estimated); Study Completion 2047-12-01 (Estimated)

PRIMARY OUTCOMES:
Liquid biopsy analyses | Day 0
  Extraction of circulating DNA or circulating RNA followed by a tumoral cells extraction.
Standard technics of disease assessment | Week 16
  Genetic and transcriptomic explorations with immunofluorescence technique. Marking with specific markers of the tumor pathology. And enumaration of tumoral cells.
Correlation between outcome 1 and outcome 2 | year 5
  Building a biological collection of blood samples and following, diagnosis and prediction of adult solid cancer.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service de Pneumologie Hôpital Louis Pradel / Groupement Hospitalier Est, Bron
  - Service de Pneumologie Hôpital Croix-Rousse / Groupement Hospitalier Nord, Lyon
  - Service de Pneumologie Aigue Spécialisée et Cancérologie Thoracique Hôpital Lyon-Sud / Groupement Hospitalier Sud, Pierre-Bénite
  - Oncologie médicale Hôpital Lyon-Sud / Groupement Hospitalier Sud, Pierre-Bénite
  - Service de dermatologie Hôpital Lyon-Sud / Groupement Hospitalier Sud, Pierre-Bénite